CLINICAL TRIAL: NCT04261166
Title: A Phase I Open Label Study to Assess the Single Dose Pharmacokinetics and Safety of Sublingual Administration of Tablets and Medicated Drops of Plant Cannabis Extract
Brief Title: A Phase I Open Label Study to Assess PK and Safety of Plant Cannabis Extract
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Breath of Life International Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BOL-PK-ST-02
Record Dates: First submitted 2020-02-04; First posted 2020-02-07 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Healthy
MeSH Terms: interventions — Dronabinol; L 644711

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Single dose (Experimental): Single dose in fasted state of : A1, A2,A3, A4, A5, B1, B2, B3, B4
  Interventions: Drug: A1; Drug: A2; Drug: A3; Drug: A4; Drug: A5; Drug: B1; Drug: B2; Drug: B3; Drug: B4
- Cross-Over food effect (Experimental): 2 doses: fasted and fed state with the same product: A1, A4, A5, B4
  Interventions: Drug: A1; Drug: A4; Drug: A5; Drug: B4
- Cross-Over product comparison (Experimental): 2 doses: in fasted state comparing A1 to A4
  Interventions: Drug: A1; Drug: A4
- Cross-over route of administration comparison (Experimental): 2 doses: in fasted state comparing oral administration to sublingual administration of A4
  Interventions: Drug: A4

INTERVENTIONS:
Drug: A1 — Medical Cannabis oil diluted in Olive oil. CBD 36.6 mg, THC 1.8 mg (6 drops)
  Other Names: Celixir 20 T1/C20- CBD 20%, THC 1%
  Arms: Cross-Over food effect; Cross-Over product comparison; Single dose
Drug: A2 — Medical Cannabis oil diluted in Olive oil. CBD 0.6 mg, THC 3.1 mg (1 drop)
  Other Names: Telixir 10 T2/C10 - CBD 2%, THC 10%
  Arms: Single dose
Drug: A3 — Medical Cannabis oil diluted in Olive oil. CBD 3.1 mg. THC 3.1 mg (1 drop)
  Other Names: Equatir 10 T10/C10 - CBD 10%, THC 10%
  Arms: Single dose
Drug: A4 — Medical Cannabis (oil diluted in MCT oil). CBD 34.8 mg, THC 1.7 mg (6 drops)
  Other Names: C18T0.9 in MCT oil - CBD 18%, THC 0.9%
Drug: A5 — Medical Cannabis oil (diluted in MCT oil). CBD 0.6 mg, THC 3.1 mg (1 drop)
  Other Names: T10/C2 - CBD 2%, THC 10%
  Arms: Cross-Over food effect; Single dose
Drug: B1 — Sublingual tablets. CBD 40 mg, THC 2 mg (1 tablet)
  Other Names: Tablet: CBD 40 mg, THC 2 mg
  Arms: Single dose
Drug: B2 — Sublingual tablets. CBD 30 mg, THC 5 mg (1 tablet)
  Other Names: Tablet: CBD 30 mg, THC 5 mg
  Arms: Single dose
Drug: B3 — Sublingual tablets. CBD 40 mg (1 tablet)
  Other Names: Tablet: CBD 40 mg
  Arms: Single dose
Drug: B4 — Sublingual tablets. CBD 40 mg (1 tablet)
  Other Names: Tablet: CBD 40 mg
  Arms: Cross-Over food effect; Single dose

SUMMARY:
This study is an open-label, single-dose, healthy volunteer phase 1 study after overnight fasting designed to study the safety and PK of medicated drops and tablet formulation for sublingual administration.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, male or female, between 18 and 45 years of age (inclusive).
2. Body mass index (BMI) between 20-30 kg/m2 (both inclusive)
3. No recent cannabis usage within 30 days from screening
4. Normal rage hepatic functions
5. No electrolytes abnormalities
6. Vital signs at screening (after five minutes resting measured in the supine position) within the following ranges:

   1. Body temperature between 35.0 to 37.5 °C
   2. Systolic blood pressure, 90 to 150 mmHg*
   3. Diastolic blood pressure, 60 to 90 mmHg*
   4. Pulse rate, 50 to 90 beats per minute*.
   5. *Blood pressure and pulse rate will be taken again in a standing position. After two minutes standing, there shall be no more than a 20 mmHg drop in systolic or 10 mmHg drop in diastolic blood pressure, associated with clinical manifestation of postural hypotension).

Exclusion Criteria:

1. Blood donation within 90 days
2. History of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastroenterology, endocrine, immunology, dermatologic, neurologic or psychiatric disorders
3. Subjects with a history of alcohol, drug abuse, chronic cannabis use within 2 years of study
4. Pregnant women
5. Subjects who used any prescription or OTC medication in the past 14 days with the exception of paracetamol or ibuprofen.
6. Sexually active males whose partner is of childbearing potential who do not agree to practice two highly effective methods of birth control or remain abstinent during the study and for three months after the last dose of IMP. Sexually active females of childbearing potential who do not agree to practice two highly effective methods of birth control or remain abstinent during the study and for three months after the last dose of IMP
7. Pregnant, lactating or planning pregnancy during the course of the study and for three months thereafter.
8. Subjects who had postural drop of > 20 mmHg in systolic blood pressure at screening
9. Patients with heart failure,
10. Subjects with a history of psychotic state in the past or anxiety disorder,
11. Subjects at age of less than 30 years with a history of psychiatric disease in a first-degree family member
12. Subjects with a history of addiction or drug abuse

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic analysis of Cmax | 0-12 hours post dose
Pharmacokinetic analysis of Tlag | 0-12 hours post dose
Pharmacokinetic analysis of Tmax | 0-12 hours post dose
Pharmacokinetic analysis of AUC(0-t) | 0-12 hours post dose
Pharmacokinetic analysis of AUC(0-∞) | 0-12 hours post dose
Pharmacokinetic analysis of %AUC extrapolated | 0-12 hours post dose
Pharmacokinetic analysis of T1/2 | 0-12 hours post dose
Pharmacokinetic analysis of clearance from plasma (Cl/F) | 0-12 hours post dose
Pharmacokinetic analysis of ratio of the Volume of distribution based on the terminal phase to the bioavailability (Vz/F) | 0-12 hours post dose
Pharmacokinetic analysis of clearance from plasma dose normalized Cmax | 0-12 hours post dose
Pharmacokinetic analysis of dose normalized AUC | 0-12 hours post dose

CONTACTS AND LOCATIONS:
Locations (1):
- Ziv Medical Center, Safed, Israel

IPD SHARING:
Plan to Share IPD: No